CLINICAL TRIAL: NCT06306066
Title: Coronary Microvascular Dysfunction in Chronic Coronary Syndrome - Invasive Assessment With Thermo-dilution Technique in the LAD and Biobanking in an All-comer Population
Brief Title: Coronary Thermo-dilution Derived Flow-indices in Chronic Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Jonas Persson, Senior Consultant, MD, PhD, Karolinska Institutet
Other Study IDs: 2015/962-31
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Microvascular Angina; Coronary Microvascular Dysfunction
Keywords: coronary microvascular dysfunction; microvascular angina; coronary artery disease; microcirculation; index of microcirculatory dysfunction; coronary flow reserve; baseline resistance index
MeSH Terms: conditions — Coronary Artery Disease; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples and whole blood obtained at index coronary angiography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
Patients scheduled for elective coronary angiography due to chronic coronary syndrome are recruited at admission to hospital before the coronary anatomy is known. Immediately after coronary angiography measures thermo-dilution derived flow indices are obtained in the left left anterior descending artery (LAD). The patients are followed through telephone-calls and medical records at 1 and 2 years after inclusion and at completion of the study. The hypothesis is that elevated index of microcirculatory resistance (IMR),(>25) is associated with all-cause death, myocardial infarction (MI) and hospitalization due to congestive heart failure (CHF).

The primary analysis is the relationship between IMR and the composite outcome all-cause death, MI and hospitalization due to CHF.

DETAILED DESCRIPTION:
Patients scheduled for elective coronary angiography due to chronic coronary syndrome are recruited at admission to hospital after written informed consent has been obtained and before the coronary anatomy is known. Blood sampling is performed from the arterial sheath before coronary angiography. The coronary angiography is done according to clinical practice. Immediately after coronary angiography measures thermo-dilution derived flow indices are obtained in the LAD (methods below). Interventions of epicardial lesions are then performed at the percutaneous coronary intervention (PCI)-operators discretion.

Fractional Flow Reserve (FFR), Coronary Flow Reserve(CFR) and IMR measurements

All indices FFR, CFR and IMR are measured in the left anterior descending artery (LAD). The flow measurements shall be obtained before PCI in the LAD. Further assessment of flow in LAD after PCI are optional. Flow measurements in the right coronary artery and circumflex lesions are optional.

Flow measurements:

A coronary guidewire with pressure and temperature sensors (PressurewireX, Abbott Inc, Calif., USA) is advanced in the LAD. The thermistor is placed > 70 mm from the catheter-tip and three millilitres of cold saline is injected into the LAD three times through the guiding catheter and thermo-dilution resting curves in triplicate are obtained. The patient then receives an intravenous infusion of adenosine (167 µg/kg/min) during approximately two minutes to induce stable hyperaemia. Again, three millilitres of cold saline is injected into the LAD through the guiding catheter and hyperaemic thermos-dilution curves in triplicate are obtained.

FFR is calculated as the ratio of distal coronary pressure (Pd) to proximal coronary pressure (Pa) at hyperaemia. CFR will be calculated through as the ratio of mean transit time of resting thermo-dilution curves (Tmnbas) divided by mean transit time of hyperaemic thermos-dilution curves (Tmnhyp). IMR is calculated as the product of Pd and Tmnhyp during stable hyperaemia. If FFR is <0.75 IMR can be overestimated and will be calculated differently (Yong et al.); Corrected index of microcirculatory resistance (IMRcorr) = Pa x Tmnhyp x ([1.35 x Pd/Pa] - 0.32).

Recordings of systolic blood pressure, diastolic blood pressure, Tmnbas, Tmnhyp, Pa, Pd, IMR, CFR will be saved and analysed off-line by a dedicated physician.

Follow-up The patients are followed through telephone-calls and medical records at 1 and 2 years and after inclusion and at completion of the study December 2022.

Patients with extensive atherosclerotic disease in the left main or the LAD with risk of complications when advancing a pressure wire making flow-measures not possible will be followed according to the protocol but excluded from the primary analysis. Patients with chronic total occlusions (CTO) in the LAD making flow-measures impossible in the LAD will be followed according to the protocol but excluded from the primary analysis.

Survival analysis The null hypothesis is that subjects with IMR >25 have the same outcome (death, MI, and hospitalization due to CHF) as subjects with IMR≤25. Assumptions are that 30% of subjects have IMR >25, the hazard ratio is 2.0, the event rate is 0.09 per year, censoring rate 0.3/year, average follow-up 3 years. With 395 subjects the power is 80% to reject the null hypothesis. α=0.05.

Biomarkers in relation to IMR Post-hoc power calculation; the null hypothesis is that no variables are associated with IMR. Assumptions; effect-size (R2) = 0.20; maximum variables in the regression analysis = 15; α = 0.05. With a power of 0.80 a sample size of 89 subjects are needed to reject the null hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stable angina pectoris or suspected angina pectoris who are scheduled for coronary angiography
* Age 18 years - 85 years
* Life expectancy >2 years

Exclusion Criteria:

* Acute coronary syndrome (ST-elevation myocardial infarction [STEMI], non-ST-elevation myocardial infarction [NSTEMI] and unstable angina pectoris)
* Known CHF
* Prior heart transplantation
* Prior coronary artery by-pass grafting
* Hypertrophic cardiomyopathy (Septum >15 mm)
* Valvular disease
* Not eligible for coronary angiogram
* Cancer within three years of admission
* Peri-myocarditis
* Atrial fibrillation with heart beats per minute >120
* Asthma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with stable angina pectoris or suspected angina pectoris who are scheduled for coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality, MI and/or hospitalization due to CHF | Study completion, approximately 5 years
  Cumulative rate of all-cause mortality, MI and/or hospitalization due to CHF at study completion

SECONDARY OUTCOMES:
Rate of all-cause mortality | Study completion, approximately 5 years
  Cumulative rate of all-cause at study completion
Rate of hospitalization due to CHF. | Study completion, approximately 5 years
  Cumulative rate of hospitalization due to CHF at study completion
Rate of all-cause mortality and/or MI | Study completion, approximately 5 years
  Cumulative rate of all-cause mortality and MI at study completion
Rate of MI | Study completion, approximately 5 years
  Cumulative rate of MI at study completion
Rate of stroke | Study completion, approximately 5 years
  Cumulative rate of Stroke at study completion
Rate of ischemic stroke | Study completion, approximately 5 years
  Cumulative rate of Ischemic stroke at study completion
Rate of unscheduled revascularization | Study completion, approximately 5 years
  Cumulative rate of Unscheduled revascularization at study completion

CONTACTS AND LOCATIONS:
Overall Officials: JONAS PERSSON, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd University Hospital and Karolinska Institutet Danderyds University Hospital (KI DS), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Murthy VL, Naya M, Foster CR, Gaber M, Hainer J, Klein J, Dorbala S, Blankstein R, Di Carli MF. Association between coronary vascular dysfunction and cardiac mortality in patients with and without diabetes mellitus. Circulation. 2012 Oct 9;126(15):1858-68. doi: 10.1161/CIRCULATIONAHA.112.120402. Epub 2012 Aug 23. PMID 22919001
- [Background] Ong P, Camici PG, Beltrame JF, Crea F, Shimokawa H, Sechtem U, Kaski JC, Bairey Merz CN; Coronary Vasomotion Disorders International Study Group (COVADIS). International standardization of diagnostic criteria for microvascular angina. Int J Cardiol. 2018 Jan 1;250:16-20. doi: 10.1016/j.ijcard.2017.08.068. Epub 2017 Sep 8. PMID 29031990
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] van de Hoef TP, Bax M, Damman P, Delewi R, Hassell ME, Piek MA, Chamuleau SA, Voskuil M, van Eck-Smit BL, Verberne HJ, Henriques JP, Koch KT, de Winter RJ, Tijssen JG, Piek JJ, Meuwissen M. Impaired Coronary Autoregulation Is Associated With Long-term Fatal Events in Patients With Stable Coronary Artery Disease. Circ Cardiovasc Interv. 2013 Aug;6(4):329-35. doi: 10.1161/CIRCINTERVENTIONS.113.000378. Epub 2013 Jul 30. PMID 23899871
- [Background] Lee JM, Jung JH, Hwang D, Park J, Fan Y, Na SH, Doh JH, Nam CW, Shin ES, Koo BK. Coronary Flow Reserve and Microcirculatory Resistance in Patients With Intermediate Coronary Stenosis. J Am Coll Cardiol. 2016 Mar 15;67(10):1158-1169. doi: 10.1016/j.jacc.2015.12.053. PMID 26965536
- [Background] Crea F, Bairey Merz CN, Beltrame JF, Kaski JC, Ogawa H, Ong P, Sechtem U, Shimokawa H, Camici PG; Coronary Vasomotion Disorders International Study Group (COVADIS). The parallel tales of microvascular angina and heart failure with preserved ejection fraction: a paradigm shift. Eur Heart J. 2017 Feb 14;38(7):473-477. doi: 10.1093/eurheartj/ehw461. No abstract available. PMID 27907892
- [Background] Ostlund-Papadogeorgos N, Ekenback C, Jokhaji F, Mir-Akbari H, Witt N, Jernberg T, Wallen H, Linder R, Tornerud M, Samad BA, Persson J. Blood haemoglobin, renal insufficiency, fractional flow reserve and plasma NT-proBNP is associated with index of microcirculatory resistance in chronic coronary syndrome. Int J Cardiol. 2020 Oct 15;317:1-6. doi: 10.1016/j.ijcard.2020.05.037. Epub 2020 May 25. PMID 32464253
- [Background] Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, Prescott E. Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J. 2012 Mar;33(6):734-44. doi: 10.1093/eurheartj/ehr331. Epub 2011 Sep 11. PMID 21911339
- [Background] De Bruyne B, Pijls NH, Smith L, Wievegg M, Heyndrickx GR. Coronary thermodilution to assess flow reserve: experimental validation. Circulation. 2001 Oct 23;104(17):2003-6. doi: 10.1161/hc4201.099223. PMID 11673336
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Aarnoudse W, Fearon WF, Manoharan G, Geven M, van de Vosse F, Rutten M, De Bruyne B, Pijls NH. Epicardial stenosis severity does not affect minimal microcirculatory resistance. Circulation. 2004 Oct 12;110(15):2137-42. doi: 10.1161/01.CIR.0000143893.18451.0E. Epub 2004 Oct 4. PMID 15466646
- [Background] Fearon WF, Aarnoudse W, Pijls NH, De Bruyne B, Balsam LB, Cooke DT, Robbins RC, Fitzgerald PJ, Yeung AC, Yock PG. Microvascular resistance is not influenced by epicardial coronary artery stenosis severity: experimental validation. Circulation. 2004 May 18;109(19):2269-72. doi: 10.1161/01.CIR.0000128669.99355.CB. Epub 2004 May 10. PMID 15136503
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Yong AS, Layland J, Fearon WF, Ho M, Shah MG, Daniels D, Whitbourn R, Macisaac A, Kritharides L, Wilson A, Ng MK. Calculation of the index of microcirculatory resistance without coronary wedge pressure measurement in the presence of epicardial stenosis. JACC Cardiovasc Interv. 2013 Jan;6(1):53-8. doi: 10.1016/j.jcin.2012.08.019. PMID 23347861
- [Derived] Shekarestan S, Jokhaji F, Ekenback C, Tornerud M, Lorstad S, Ljungman P, Ostlund-Papadogeorgos N, Linder R, Samad B, Persson J. Elevated Resting Coronary Blood Flow Is Associated With Death, MI, and HF in All-Comer Patients With Chronic Coronary Syndrome. Circ Cardiovasc Interv. 2026 Jan 15:e015867. doi: 10.1161/CIRCINTERVENTIONS.125.015867. Online ahead of print. PMID 41537270